CLINICAL TRIAL: NCT02854982
Title: Impact on Quality of Life 3 Years After Diagnosis of Prostate Cancer
Acronym: EPICAP-QALY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LIGUE/2014/NH-001
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2018-08

CONDITIONS: Prostatic Neoplasms; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prostate Cancer: Group drawn of the case group of the case control study, entitled EPICAP
  Interventions: Procedure: therapeutic management of the prostate Cancer as usual
- No Prostate Cancer: Group drawn of the control group of the case control study, entitled EPICAP

INTERVENTIONS:
Procedure: therapeutic management of the prostate Cancer as usual
  Groups: Prostate Cancer

SUMMARY:
To study the quality of life of patients with prostate cancer at a distance from their care at a time when they are supposed to have taken a "normal" life and compared to subjects without cancer prostate of the same age.

ELIGIBILITY:
- exposed group

Inclusion Criteria:

* prostate cancer diagnosed from 1 December 2011 to 31 December 2014
* under 75 and residing in the Hérault department at diagnosis
* recruited in the EPICAP study

Exclusion criteria:

* having relapsed in the range
* non-exposed group:

Inclusion Criteria:

* controls (without prostate cancer) recruited in the EPICAP study
* matched to cases on age (5 years)
* residing in the Hérault department

Exclusion criteria:

* diagnosis of prostate cancer set in the range

Max Age: 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Target population: incident cases of prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
EORTC Quality of Life Questionnaire - Core 30 Score (EORTC QLQ-C30 Score) | 3 years from diagnosis for cases of prostate cancer and from recruitment for controls

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Houede N, Rebillard X, Bouvet S, Kabani S, Fabbro-Peray P, Tretarre B, Menegaux F. Impact on quality of life 3 years after diagnosis of prostate cancer patients below 75 at diagnosis: an observational case-control study. BMC Cancer. 2020 Aug 12;20(1):757. doi: 10.1186/s12885-020-07244-y. PMID 32787797